CLINICAL TRIAL: NCT01503463
Title: Renewing Health RCT for the Evaluation of Remote Monitoring of Patients With Congestive Heart Failure (CHF) in Central Greece
Brief Title: Remote Monitoring of Patients With CHF in Central Greece
Acronym: RHCluster7GR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Regional Health Authority of Sterea & Thessaly (Other Government)
Collaborators: Ministry for Health and Social Solidarity, Greece (Other); Municipality of Trikala, Greece (Other); Institute of Biomedical Research & Technology, Larissa, Greece (Other); Institute of Communications and Computer Systems, Athens, Greece (Other); Alexander Technological Educational Institute, Thessaloniki, Greece (Other); University of Macedonia, Thessaloniki, Greece (Other); University of Thessaly (Other)
Responsible Party: Principal Investigator, Filippos Triposkiadis, Proffesor, Director of the Cardiology Department, University Hospital of Larissa, Regional Health Authority of Sterea & Thessaly
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: FR2016; EC Grant Agreement 250487 (Other Grant/Funding Number: European Commission CIP/PSP-ICT Grant Agreement 250487)
Record Dates: First submitted 2012-01-02; First posted 2012-01-04 (Estimated); Last update posted 2015-03-20 (Estimated); Status verified 2015-03

CONDITIONS: Congestive Heart Failure
Keywords: Congestive Heart Failure; Telemedicine
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Usual Care (No Intervention): Patients in the control group receive usual care delivered by their primary care physicians and cardiologists. Usual care consists of regular visits to the specialist or primary care clinics every time a medication change is required, or a medical examination is needed.
- Home telemonitoring of patients with CHF (Experimental)
  Interventions: Procedure: Home telemonitoring of patients with CHF

INTERVENTIONS:
Procedure: Home telemonitoring of patients with CHF — Patients in the intervention group receive a personal 1-lead or 12-lead ECG recorder, a blood pressure monitor, a digital weight scale and appropriate education regarding the use of these devices. ThA trained nurse visits the patients weekly during the first month, and monthly thereafter, to confirm the appropriate use of the devices and services, to monitor symptoms, adherence to pharmacological and non-pharmacological treatment, and to complete the case record forms when necessary.
  If there is deterioration in the monitored vital signs, or if symptoms are reported, the allocated cardiologist is informed via the telehealth platform and has to decide whether the patient has to visit the hospital as in- or outpatient and whether the therapy has to be modified.
  Arms: Home telemonitoring of patients with CHF

SUMMARY:
The purpose of this study is to evaluate whether telemonitoring of patients with chronic heart failure produces a reduction in the combined end point of all cause mortality and number of hospitalisations, and whether it improves health related quality of life. In addition, the trials evaluate the economic and organisational impact of the telemonitoring service and examine its acceptability by patients and health professionals.

DETAILED DESCRIPTION:
The purpose of this study is to the evaluate the use of a mobile and PSTN phone-based telehealth platform will be able to produce a reduction in the combined end point of all cause mortality, will have positive or negative impact in their generic and disease specific quality of life , or their specific activity compared with usual care. Following this; it is also hypothesized that this will also lead to a change in overall risk for CHF complications. In addition the patients' satisfaction using the telemedicine service will be studied. A Cost-Effective Analysis and Cost Utility Analysis will evaluate the tele-health service compared with the usual care from the health and social perspective.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 65 years.
* Discharge from hospital after acute heart failure in the previous 3 months and FE < 40% or FE > 40% plus BNP > 400 (or plus NT-proBNP>1500) during hospitalization

Exclusion Criteria:

* Comorbidities prevalent on CHF with life expectation < 12 months.
* Inability to use the equipment and help at home not available.
* Myocardial infarction or percutaneous coronary intervention in the last 3 months.
* Coronary artery bypass, valve substitution or correction in the last 6 months or scheduled.
* Being on waiting list for heart transplantation.
* Being enrolled in other trial.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-03; Primary Completion 2013-12 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Combined end point of all cause mortality | 12 months minimum
Number of hospitalisations for heart failure | 12 months minimum

SECONDARY OUTCOMES:
Cardiovascular and all-cause mortality | 12 months minimum
Health related quality of life as measured by the SF-36 v2 | 12 months minimum- at the entry point of the intervention and the end
Patient's specific activity using Specific activity questionnaire (SAQ) and the Veterans specific activity questionnaire (VSAQ) | 12 months minimum- at the entry point of the intervention and the end.
Disease Specific Quality of Life using the Minnesota Living with Heart Failure questionnaire (MLHF) | 12 months minimum- at the entry point of the intervention and the end.
Economic Evaluation (Cost-Effective Analysis- Cost Utility Analysis) | 12 months minimum
Patients' Acceptance-Satisfaction measured by the WSD Questionnaire | at 2nd and at 12th month

CONTACTS AND LOCATIONS:
Overall Officials: Filippos Triposkiadis, MD, PhD, Principal Investigator — Cardiology Department - Regional University Hospital of Larisa
Locations (1):
- Cardiology Department - Regional University Hospital of Larisa, Larissa, Thessaly, Greece

REFERENCES:
- [Background] Scherr D, Kastner P, Kollmann A, Hallas A, Auer J, Krappinger H, Schuchlenz H, Stark G, Grander W, Jakl G, Schreier G, Fruhwald FM; MOBITEL Investigators. Effect of home-based telemonitoring using mobile phone technology on the outcome of heart failure patients after an episode of acute decompensation: randomized controlled trial. J Med Internet Res. 2009 Aug 17;11(3):e34. doi: 10.2196/jmir.1252. PMID 19687005
- [Background] Clark RA, Inglis SC, McAlister FA, Cleland JG, Stewart S. Telemonitoring or structured telephone support programmes for patients with chronic heart failure: systematic review and meta-analysis. BMJ. 2007 May 5;334(7600):942. doi: 10.1136/bmj.39156.536968.55. Epub 2007 Apr 10. PMID 17426062
- [Background] Cleland JG, Louis AA, Rigby AS, Janssens U, Balk AH; TEN-HMS Investigators. Noninvasive home telemonitoring for patients with heart failure at high risk of recurrent admission and death: the Trans-European Network-Home-Care Management System (TEN-HMS) study. J Am Coll Cardiol. 2005 May 17;45(10):1654-64. doi: 10.1016/j.jacc.2005.01.050. Epub 2005 Apr 22. PMID 15893183
- [Background] Klersy C, De Silvestri A, Gabutti G, Regoli F, Auricchio A. A meta-analysis of remote monitoring of heart failure patients. J Am Coll Cardiol. 2009 Oct 27;54(18):1683-94. doi: 10.1016/j.jacc.2009.08.017. PMID 19850208
- [Background] Inglis SC, Clark RA, McAlister FA, Ball J, Lewinter C, Cullington D, Stewart S, Cleland JG. Structured telephone support or telemonitoring programmes for patients with chronic heart failure. Cochrane Database Syst Rev. 2010 Aug 4;(8):CD007228. doi: 10.1002/14651858.CD007228.pub2. PMID 20687083
- [Background] Inglis SC, Clark RA, McAlister FA, Stewart S, Cleland JG. Which components of heart failure programmes are effective? A systematic review and meta-analysis of the outcomes of structured telephone support or telemonitoring as the primary component of chronic heart failure management in 8323 patients: Abridged Cochrane Review. Eur J Heart Fail. 2011 Sep;13(9):1028-40. doi: 10.1093/eurjhf/hfr039. Epub 2011 Jul 6. PMID 21733889
- [Background] Chaudhry SI, Mattera JA, Curtis JP, Spertus JA, Herrin J, Lin Z, Phillips CO, Hodshon BV, Cooper LS, Krumholz HM. Telemonitoring in patients with heart failure. N Engl J Med. 2010 Dec 9;363(24):2301-9. doi: 10.1056/NEJMoa1010029. Epub 2010 Nov 16. PMID 21080835
- See also: "The Renewing Health project is partially funded under the ICT Policy Support Programme (ICT PSP) as part of the Competitiveness and Innovation Framework Programme by the European Community" — http://www.renewinghealth.eu/